CLINICAL TRIAL: NCT07355426
Title: Pediatric In-Hospital Mortality Risk in Congolese Children With Severe Malaria: Derivation of Clinical Prediction Models Using Machine Learning Based-Algorithms
Brief Title: Clinical Prediction Models for Pediatric In-Hospital Death Risk in Congolese Severe Malaria Children Using Machine Learning Based-Algorithms
Status: Completed | Type: Observational
Sponsor: University of Kinshasa (Other)
Responsible Party: Principal Investigator, Ken Bisabu, Kelu, Principal Investigator, University of Kinshasa
Other Study IDs: SM_PEDCUK
Record Dates: First submitted 2025-09-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Severe Malaria
Keywords: Severe malaria; Paediatric in-hospital mortality risk; Machine learning-based algorithms; Predictive model; Plasmodium falciparum; Multiple Organ Dysfunction Syndrome (MODS); Metabolic acidosis
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Multiple Organ Failure; Acidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples Without DNA — Arterial blood sample and one-drop finger pulp blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEDCUK_0000: Children aged 2 to 9 years, admitted to the paediatric intensive care units for severe malaria
  Interventions: Diagnostic Test: Puncture of the radial artery for instant arterial blood gaz as well as for venous biochemistry

INTERVENTIONS:
Diagnostic Test: Puncture of the radial artery for instant arterial blood gaz as well as for venous biochemistry — 1. The puncture of the radial artery was made for the instant arterial blood gaz as well as for venous biochemistry
  2. The one-drop finger pulp blood test was made for parasitemia measurement and the rapid diagnosis test for plasmodium falciparum

SUMMARY:
The goal of this observational study is to optimize the management of severe childhood malaria, based on understanding and controlling the severity factors of the disease in Congolese children aged 2 to 9 years (the age group at risk of developing various severe forms of malaria), admitted to the paediatric intensive care units (PICU).

The main question it aims to answer is whether the scores or models used to predict the severity of severe malaria and the associated risk of mortality accurate enough to warrant early interventions, including treatments, on their own?

Thus, investigators aim to fill three knowledge gaps associated with the following hypotheses:

Hypothesis-1: Children with severe malaria show signs of disease severity based on their severity scores on admission. Higher severity scores on admission are associated with a higher risk of mortality.

Hypothesis-2: Validation of the predictive power and transferability of severe malaria severity scores to additional independent populations is needed to support their clinical utility.

Hypothesis-3: The severity of the clinical and biological changes induced by plasmodium depends not only on the ability of the parasite to invade and grow in the host organism, but also and above all on the number of parasites present in the host (parasitemia).

For any child admitted to the PICU and meeting the inclusion criteria, as part of clinical care, investigators proceeded before any treatment:

1. An arterial blood sample of 3 ml by puncture of the radial artery for instant arterial blood gaz as well as for venous biochemistry, including albumin, phosphate, chlorine, magnesium, urea, creatinine and total bilirubin dosages, and,
2. A one-drop finger pulp blood test for parasitemia measurement and the rapid diagnosis test for plasmodium falciparum.

Then, the diagnostic parameters of acid-base disorders will be calculated, including AG (anion gap), AGCAP (AG corrected for albumin and phosphate plasmatic concentrations), SIG (Strong ion gap), SBE (Standard base excess) and SBDCAP (Standard base deficit corrected for albumin and phosphate plasmatic concentrations).

DETAILED DESCRIPTION:
Background:

Severe malaria has associated with a high risk of paediatric hospital mortality in resource-constrained countries, which remains deplorable. Improved methods of risk-stratification can assist in referral decision making and resource allocation. Investigators aim to i) create prediction model for in-hospital mortality risk among children presenting with severe malaria and compare its predictive performance to the current models, ii) validate the latter, and iii) assess the plasmodium-induced changes in clinical and biological parameters.

Methods:

This is a retrospective study of data collected prospectively during a period from January 30, 2017 to August 01, 2025, from children with severe malaria, admitted to the PICU of the Monkole Hospital Center (MHC) and the Kimbondo Pediatric Center (KPC), all in Kinshasa, DR. Congo. Baseline clinical and laboratory variables were collected on enrolled children. The primary outcome is death up to 1 week post-admission, and the second outcome, the length of stay in pediatric intensive care following admission for severe malaria. Machine learning algorithms will be employed to accomplish the three specific research objectives.

Expected Results:

In line with research objectives, the following results are expected:

1. The prevalence of Multiple Organ Dysfunction Syndrome (MODS) and metabolic acidosis in children presenting with severe malaria will be determined.
2. A novel model for predicting associated mortality risk of severe malaria will be developed:

   1. This novel model will be based on predictors of disease severity and will measure:

      * The degree of severity of MODS and metabolic acidosis.
      * The length of stay for severe malaria in the PICU
      * The risk of death following hospitalization for severe malaria
      * The influence of parasitemia on disease severity
   2. The performance of the proposed novel model will be measured
   3. The predictive nomogram and scoring system will be associated with it.
3. Investigators validate and compare the performance of existing models for predicting severe malaria severity against the proposed novel model.

Together, research data will provide proof of principle supporting early interventions and treatment choices in children presenting with severe malaria.

ELIGIBILITY:
I) Inclusion Criteria:

-Admission to the pediatric intensive care unit (PICU) for severe malaria, as defined by the World Health Organization (WHO) criteria.

Definitions:

1. Severe malaria was defined by the presence of at least one major clinical manifestation, including:

   * Coma
   * Repeated seizures (≥ 2 episodes within 24 hours)
   * Neurological disorders
   * Respiratory distress
   * Liver failure
   * Dark ("Coca-Cola") urine
   * Jaundice
   * Renal failure (anuria)
   * Severe anaemia (Hb ≤ 5 g/dL)
   * Bleeding abnormalities
   * Circulatory collapse or systolic blood pressure < 50 mmHg
2. Data collection periods varied by health zone and clinical unit. However, within each zone, all consecutively admitted patients during the study period were included.

II) Exclusion Criteria:

* Another medical condition (non-parasitic infection or other) capable of causing anemia or similar abnormalities.
* Comorbidities that could interfere with the clinical presentation or outcomes of severe malaria.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with severe malaria, admitted to the pediatric intensive care units of the Monkole Hospital Center (MHC) and the Kimbondo Pediatric Center (KPC), all in Kinshasa, DR. Congo.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is death during hospitalization for severe malaria [From day 1 of admission to the pediatric intensive care unit (PICU) up to day 7 post-admission] | Day 7
  Death was defined as a categorical variable, defining patients who died and those who survived.

SECONDARY OUTCOMES:
The secondary outcome is survival time, defined as the interval between hospital admission and death occurring during the hospitalization period [From day1 of admission until death/recovery (discharge from hospital), assessed up to day7 post-admission] | From day 1 of admission to the PICU until death or recovery (discharge from hospital), assessed up to day 7 post-admission.
  Survival Time was defined as the interval between hospital admission for severe malaria and death occurring during the hospitalization period. The hospitalization period extended from day 1 of admission to death (for non-survivors) or discharge (for survivors). Patients who were still alive at the end of the hospitalization period of up to day 7 (follow-up period for each patient = 7 days) or those lost to follow-up were considered censored.

CONTACTS AND LOCATIONS:
Overall Officials: Celestin Ndosimao Nsibu, Full professor, Study Director — Kinshasa University; Joseph Mabiala Bodi, Full professor, Study Chair — Kinshasa University; Leon Tshilolo, Full professor, Study Chair — Kinshasa University
Locations (1):
- Kinshasa, Kinshasa, Kinshasa City, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berkley JA, Ross A, Mwangi I, Osier FH, Mohammed M, Shebbe M, Lowe BS, Marsh K, Newton CR. Prognostic indicators of early and late death in children admitted to district hospital in Kenya: cohort study. BMJ. 2003 Feb 15;326(7385):361. doi: 10.1136/bmj.326.7385.361. PMID 12586667
- [Background] Kumar N, Thomas N, Singhal D, Puliyel JM, Sreenivas V. Triage score for severity of illness. Indian Pediatr. 2003 Mar;40(3):204-10. PMID 12657751
- [Background] Helbok R, Kendjo E, Issifou S, Lackner P, Newton CR, Kombila M, Agbenyega T, Bojang K, Dietz K, Schmutzhard E, Kremsner PG. The Lambarene Organ Dysfunction Score (LODS) is a simple clinical predictor of fatal malaria in African children. J Infect Dis. 2009 Dec 15;200(12):1834-41. doi: 10.1086/648409. PMID 19911989
- [Background] Njim T, Tanyitiku BS. Prognostic models for the clinical management of malaria and its complications: a systematic review. BMJ Open. 2019 Nov 26;9(11):e030793. doi: 10.1136/bmjopen-2019-030793. PMID 31772089
- [Background] World malaria report 2024. Geneva: World Health Organization. 2024

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT07355426/Prot_SAP_000.pdf